CLINICAL TRIAL: NCT04185233
Title: Comparison in Anxiety and Pain Scores Between Distraction and Nitrous Oxide for Procedural Pain in Children Aged 3 to 9 Years : a Randomized Clinical Trial
Brief Title: Distraction and Nitrous Oxide for Venous Puncture
Acronym: DISPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Walid HABRE, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: in progress
Record Dates: First submitted 2019-05-09; First posted 2019-12-04 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Anxiety; Pain; Venous Puncture
Keywords: nitrous oxide; distraction
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPad distraction (Experimental): Children of this group will receive the iPad when the nurse will prepare the material for the venous track. They will choose a game adapted to their age and will be able to play it during all the procedure time.
  Intervention : game on iPad
  Interventions: Other: Games on an iPad
- Nitrous Oxide (Active Comparator): Children of this group will receive the Nitrous Oxide 3 minutes before the intervention (venous track). They will keep the mask during all the procedure time.
  Intervention : Nitrous Oxide
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Other: Games on an iPad — Many games will be programmed on the iPad and organized by age. The child will choose one game and play it during all the procedure time.
  Arms: iPad distraction
Drug: Nitrous Oxide — Nitrous oxide will be provided to the child by a mask 3 minutes before the intervention and during all this one.
  Arms: Nitrous Oxide

SUMMARY:
This study will compare the efficiency of the iPad distraction or the administration of Nitrous Oxide on the anxiety decrease when a peripheral venous catheter is needed in children between 3 and 9 years old.

DETAILED DESCRIPTION:
The study is aiming at demonstrating the efficacy of active distraction by an iPad on the anxiety consequent to venipuncture and insertion of a peripheral vein catheter. The comparator is nitrous oxide in a 50% mixture with oxygen that is routinely used for sedation during procedural pain. However, nitrous oxide has secondary effects particularly on the inhibition of Vitamin B12.

The primary outcome is anxiety scores. Secondary outcomes are pain scores and satisfaction of parents and health providers.

All children will have EMLA cream (mixture prilocaine and lidocaine) applied one hour prior to venous punction. Anxiety, pain and satisfaction scores will be recorded at baseline and then within an hour following the venipuncture and insertion of the peripheral vein catheter.

ELIGIBILITY:
Inclusion Criteria:

* Venous track needed
* French mother tongue
* Age between 3 and 9 years old

Exclusion Criteria:

* Children with cognitive disorder (autism, metabolic disorders,
* Children with cerebral-motor disability
* Children who don't speak french
* Children with ADHD treatment
* Children with epilepsy
* Children who present contraindication to the use of Nitrous oxide

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Anxiety score | From one hour prior to venous puncture until 1 hour afterwards
  Anxiety level measured by a scale (modified Yale Preoperative Anxiety Scale) measured at baseline, during the venous puncture and one hour afterwards. The scale scores from a minimum of 5 (no anxiety) to 22 (extremely anxious).

SECONDARY OUTCOMES:
Pain score | From one hour prior to venous puncture until 1 hour afterwards
  Pain intensity level will be measured at baseline, during the venous puncture and one hour afterwards, by a scale (Visual analog scale), which includes a score of 0 (no Pain) to 10 (worse pain).

OTHER OUTCOMES:
Satisfaction score | From time of venous puncture until 1 hour afterwards
  Satisfaction of parents and care givers about the cares given to the child using a rating scale from 1(not satisfied at all) to 10 (extremely satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Manon Cadoux, Student, Principal Investigator — University of Geneva; Virginie Luscher, Student, Principal Investigator — University of Geneva
Locations (1):
- Geneva Children's Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided